CLINICAL TRIAL: NCT06620276
Title: Acceptance and Commitment Therapy in Patients With Alcohol Use Disorder and Comorbid Treatment-Resistant Depression Who Are Undergoing Ketamine Intervention: A Feasibility Study
Brief Title: ACT_for Alcohol Use Disorder and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-12519
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Depression - Major Depressive Disorder; Alcohol Use Disorder
Keywords: Depression; Psychotherapy; Alcohol Use Disorder; Ketamine-assisted Acceptance and Commitment Therapy
MeSH Terms: conditions — Alcoholism; Depression | interventions — Acceptance and Commitment Therapy; Ketamine

STUDY DESIGN:
Intervention Model Description: Assessing the feasibility of providing Acceptance and Commitment Therapy (ACT) to patients diagnosed with Alcohol Use Disorder and Treatment-Resistant Depression who are undergoing ketamine sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine-assisted Acceptance and Commitment Therapy (Experimental): 30 consecutive participants who will receive 6 infusions of ketamine and 8 sessions of Acceptance and Commitment Therapy (ACT) at our research site.
  Interventions: Behavioral: Acceptance and Commitment Therapy; Drug: Ketamine

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The ACT intervention consists of eight weekly 50 minute sessions, delivered in person when possible, with virtual options available. ACT targets psychological flexibility by addressing fusion, evaluation, avoidance, and reason giving through six core processes: acceptance, values, committed action, present moment awareness, cognitive defusion, and self as context. Sessions combine didactic content and experiential exercises following a standardized manual, with therapists trained in ACT. Participants receive a workbook to support practice. Each session begins with a brief mindfulness exercise that evolves across weeks, starting with grounding and simple emotional labeling, then progressing to neutral sensory descriptions and openness to challenging sensations.
Drug: Ketamine — The protocol includes 6 IV ketamine infusions over 4 weeks at the CHUM Neuromodulation Unit, following the Montreal Model integrating psychotherapeutic and contextual elements (e.g. preparation, music, and integration).
  Infusions occur twice weekly in weeks 3 and 4 of the treatment protocol, then once weekly in weeks 5 and 6. The first dose is 0.5 mg/kg in 250 mL saline over 40 minutes, with possible titration up to 1.0 mg/kg based on tolerability, clinical response, and participant preferences. Blood alcohol level is measured by breathalyzer before each session, and if any detectable alcohol is present (i.e., BAC ≠ 0%), the infusion will be postponed and rescheduled.
  Infusions occur in a quiet, dim room with continuous monitoring. Before each infusion, a brief mindfulness exercise promotes openness to internal experience. During the infusion, participants listen to a curated 60 minute instrumental playlist to support emotional exploration.

SUMMARY:
Alcohol use disorders (AUDs) and depressive disorders frequently coexist, complicating the clinical management of patients suffering from them.

Taken separately, these two disorders have a significant prevalence in the population, and a recent meta-analysis concluded that coexistence could reach 1 in 5 patients (20.8%). This comorbidity represents a considerable challenge, particularly in cases of treatment-resistant depression (TRD), where patients do not respond to conventional pharmacological interventions.

Since alcohol can act as a powerful trigger for depressive symptoms, and conversely, a depressive state increases the risk of alcohol abuse, the question of intervention sequence is also of clinical interest: should priority be given to treating TRD, AUD or both simultaneously? This question raises a major issue for healthcare professionals, as current conventional therapeutic approaches present limitations in the concomitant management of these complex disorders.

Thus, in certain clinical settings, ketamine has emerged as a promising intervention to treat both TRD and AUD. In fact, ketamine has been shown to produce rapid but only transient antidepressant effects, and is part of the possible treatment arsenal for TRD. The potential of ketamine in the treatment of AUD has also been explored in recent studies, with a few small randomized controlled trials. In these trials, the combination of ketamine with psychotherapy, versus placebo, was investigated as a means of alleviating AUD. Ketamine was shown to increase abstinence rates, time to relapse and decrease the number of heavy drinking days.

Acceptance and Commitment Therapy (ACT) is a form of cognitive-behavioural therapy that emphasizes psychological flexibility and acceptance of difficult emotions and thoughts without judgment, a type of psychotherapy particularly relevant to AUD. Thus, adding ACT to ketamine treatment could increase the duration of ketamine's effect on depressive symptoms, while reducing AUD.

In view of this accumulated evidence of the potential benefit of ketamine and ACT, adding acceptance and commitment therapy to ketamine appears to be a promising option for improving outcomes in patients diagnosed with TRD comorbid with AUD. This study will not only verify the feasibility of this type of intervention in this particular patient population, but also the preliminary effects on their alcohol consumption and depressive symptoms.

DETAILED DESCRIPTION:
Study rationale Acceptance and Commitment Therapy (ACT) has been proposed as a particularly well-suited form of psychotherapy to be added to ketamine for improving its rapid but short antidepressant action. This is in part because of ketamine's acute effect on psychological flexibility, a crucial construct that is addressed with ACT.

There has been extensive efforts to find effective strategies to enhance and sustain the therapeutic response of ketamine, with most attempts using various pharmacotherapies-such as clonidine, D-cycloserine, lamotrigine, lithium, rapamycin, and riluzole- which have yielded mostly disappointing results. Consequently, the most common approach to extending ketamine benefits has been to administer repeated doses, although there is limited evidence supporting the long-term safety, efficacy, and practicality of this practice.

Substantial evidence indicates that psychotherapy can enhance the effects of pharmacological treatments, such as oral antidepressants, and even help maintain their benefits after discontinuation. While further research is required, it is plausible to assume that similar benefits of adding psychotherapy could extend to ketamine, particularly considering its potential neuroplastic effects.

In view of the accumulated evidence, the addition of ACT to a ketamine intervention appears as a promising option to improve the outcomes of patients diagnosed with AUD comorbid with TRD. This study will not only verify the feasibility of adding psychotherapy to ketamine in this population, but also the effect on their alcohol consumption and depressive symptoms.

Background Alcohol Use Disorder (AUD) and depressive disorders frequently coexist and complicate the clinical management and treatment outcomes for patients. It is estimated that around 1 in 10 people (10.4%) in the USA is experiencing a major depressive disorder (MDD) in the course of a year, while it goes up to 1 in 5 (20.6%) in the course of a lifetime. As for AUD, twelve month and lifetime prevalence are respectively 13.9% and 29.1%. When these disorders coexist, the prevalence is estimated as high as 20.8%, as reported by a recent meta-analysis. Research has also shown that individuals with AUD are approximately 2.3 times more likely to experience MDD within a given year.

This comorbidity presents a formidable challenge, particularly in cases of Treatment-Resistant Depression (TRD), a subset of MDD where patients do not respond to conventional pharmacological interventions. In the United States, it is estimated that out of 8.9 million adults receiving medication for MDD, 2.8 million, or 30.9%, are grappling with TRD. The economic impact is substantial, with the total annual cost of medication-treated MDD reaching $92.7 billion, nearly half of which-$43.8 billion or 47.2%-is attributable to TRD.

The concomitance of TRD and AUD represents a major clinical challenge as alcohol can act as a powerful trigger for depressive symptoms, and conversely a depressive state can increase the risk of alcohol abuse. This creates a complex, bidirectional relationship between the two disorders, considerably complicating the assessment and clinical management of these concurrent disorders. The question of intervention sequence is also of clinical interest: should treatment of TRD, AUD, or both simultaneously be prioritized? This question raises major challenges for health professionals, as current conventional therapeutic approaches present limitations in the concomitant management of these complex disorders. Traditional pharmacological treatments, such as antidepressants, may not be sufficiently effective or tolerated by some patients to treat these comorbid disorders. As for standard psychotherapeutic approaches, such as cognitive-behavioral therapy, the heterogeneity of symptoms and diversity of issues often mean that the needs of individuals suffering from these comorbidities cannot be met comprehensively.

In response to this challenge, in selected clinical settings, ketamine has emerged as a promising intervention for treating both AUD and depressive disorders. Ketamine, an NMDA receptor antagonist, has been shown to produce rapid and substantial, albeit short-lived (i.e. 7 days), antidepressant effects in individuals with TRD. Furthermore, ketamine potential in treating AUD has been explored in recent studies, with randomized controlled trials emerging. In such trials, the combination of ketamine to psychotherapy as compared to a placebo is studied to alleviate AUD. For instance, individuals with AUD who received a ketamine infusion and motivational therapy had improved rates of abstinence, prolonged time to relapse, and fewer days of heavy drinking than individuals with AUD who received an infusion of midazolam, considered as a placebo. Another team also compared the use of ketamine with a relapse prevention-based psychological therapy to placebo and found that there was a significant increase in the number of days abstinent from alcohol.

Considering the substantial but transient effect of ketamine on depressive symptomatology, and its promising results in AUD patients, a novel approach is to add a psychotherapeutic component to the ketamine treatment with the aim of enhancing and prolonging its effect. Acceptance and Commitment Therapy (ACT) seems to be a particularly well-suited form of psychotherapy to be added to ketamine treatment. Indeed, ACT is a form of cognitive-behavioural therapy that emphasizes psychological flexibility and the acceptance of difficult emotions and thoughts without judgment. ACT has been extensively studied in various psychopathologies, including anxiety and depression, demonstrating positive outcomes in multiple rigorous clinical trials and meta-analysis. Growing evidence suggest that ACT may be an effective and even superior treatment for individuals with substance use disorders ACT encourages individuals to commit to behavior changes consistent with their values, which can be particularly beneficial for those with AUD and comorbid TRD. Ketamine has been shown to have an acute effect on psychological flexibility, and the addition of ACT's focus on acceptance and value-driven behavior holds promise for improving the ketamine's rapid and short antidepressant action and addressing the complex interplay of AUD and TRD.

Standard treatment options

Alcohol Use Disorder (AUD):

In 2023, a committee of AUD specialists published the Canadian guideline with treatment recommendations for AUD. As a strong recommendation, they first proposed that all patients with AUD should be offered specialist-led psychosocial treatment interventions, such as cognitive behavioral therapy or family-based therapy. However, both therapies were found to have small to medium beneficial impacts on AUD outcomes. For pharmacotherapy, as a complement to the psychosocial treatment, naltrexone or acamprosate were recommended as first-line therapy. Second-line options, some of them being used as off-label therapies, were also proposed, namely gabapentin, topiramate and disulfiram. Of note, these recommendations are in line with other reviews of AUD pharmacotherapy and other national guidelines (namely American and Australian guidelines).

However, there are some limitations associated with the use of those treatment options. Apart from safety concerns, with common AE associated with treatments (nausea, dizziness and fatigue, among others), there is an ongoing debate among experts about the actual efficacy of the treatment options. In fact, naltrexone and acamprosate have an estimated number needed to treat to prevent a return to heavy drinking of 12, with modest differences found when comparing drugs with placebo, contributing to their underutilization in AUD patients. For instance, in over 28,000 Medicare beneficiaries hospitalized with a primary or secondary diagnosis of AUD, it was found that only 0.7% of patients started pharmacotherapy within two days after discharge and 1.3% within 30 days. Even among patients for whom AUD was the primary diagnosis after hospitalization, only 2.3% started pharmacotherapy within two days of discharge.

Treatment Resistant Depression (TRD):

Leading experts in TRD summarized in 2023 the options available to try and reach a favorable outcome in individuals who fail to respond to at least two adequate trials of psychotropics against depression. First, extending a current antidepressant trial could be a potential treatment plan. A systematic review determined that up to 20% of patients who did not respond to their antidepressant in the first four weeks of treatment responded during the following four weeks (from weeks five to eight), and up to 10% during weeks nine to twelve. Similarly, there is some evidence, albeit conflicting, that switching antidepressants or combining antidepressants could benefit some patients, especially if the change or addition involves a new mechanism of action. To cite only one example of this option, adding antidepressants with antagonism activity on the alpha-2 receptor (i.e., mirtazapine, trazodone) to a selective serotonin reuptake inhibitor was superior to monotherapy in a meta-analysis.

Other treatment modalities have also been studied, including adding various pharmacological agents like second-generation antipsychotics and mood stabilizers. In real-world settings, most patients with TRD are prescribed multiple psychotropic medications, often for extended periods, with generally limited success. For example, a recent cohort study conducted over 12 months across various European countries, involving 411 patients with TRD, highlighted high rates of polypharmacy alongside modest clinical improvement-only about 30% showed a positive response after 6 to 12 months of consistent treatment. The study also indicated a concerning level of therapeutic inertia, where 60% of patients did not undergo any changes in their treatment plan, despite ongoing poor outcomes.

Electroconvulsive therapy (ECT), aside from the usual pharmacological approaches, is considered one of the most empirically supported interventions for TRD. However, despite its effectiveness, ECT is often hindered by significant barriers, including societal stigma, inconsistent access, and notable side effects such as memory loss, largely due to the need for general anesthesia during the procedure.

Amid the current treatment challenges, the rapid and robust antidepressant effects of subanesthetic doses of IV racemic ketamine-a distinctive N-methyl-D-aspartate (NMDA) receptor antagonist-have sparked considerable interest and optimism. Meta-analyses suggest that nearly half of patients with treatment-resistant depression (TRD) experience a significant reduction in depressive symptoms (over 50%) within just hours to days following a single 40-minute IV ketamine infusion. This promising efficacy has led many experts to regard subanesthetic ketamine as one of the most transformative advancements in psychiatric pharmacology in recent decades. While impressive, ketamine's benefits typically fade within days or weeks.

Given the evidence of ketamine's beneficial effect, the neuromodulation service of the CHUM began providing this treatment to patients with TRD in 2018, covering the whole province of Quebec. Since then, the neuromodulation service has created a state-of-the-art infrastructure for the ketamine service.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent after reading and understanding the patient information handout
* Alcohol Use Disorder (AUD) diagnosed by a trained psychiatrist
* Diagnosis of treatment resistant unipolar or bipolar depression, defined as failure to respond to ≥2 adequate trials per Canadian national depression guidelines
* Willingness to engage in 8 weekly psychotherapy sessions
* No changes to psychotropic medications during treatment
* Average daily ethanol consumption of at least moderate risk as per WHO risk levels (Men: >40 to 60 g per day or >2.9 to 4.3 drinks / Women: >20 to 40 g per day or >1.4 to 2.9 drinks)
* Bipolar or unipolar depressive episode (DSM5), current episode, with MADRS ≥ 20
* Age 18 to 70 years
* Agreement to abstain from consuming grapefruit juice on ketamine infusion days
* Agreement to abstain from driving or operating heavy machinery after infusions until the next day

Exclusion Criteria:

* Current participation in other evidence based psychotherapeutic interventions for mood disorders or substance abuse
* Inability to commit to the study protocol due to professional or personal obligations
* Non English or non French speaking
* Psychiatric comorbidity likely to take precedence over AUD or TRD
* Acute psychotic disorder or acute psychotic symptoms
* Current or prior substance abuse or dependence other than AUD (except caffeine or nicotine)
* Non response to esketamine or ketamine during the current depressive episode
* Known intellectual disability or autism spectrum disorder
* Inability to attend regular visits to the CHUM Neuromodulation clinic
* Depression secondary to stroke, cancer, or severe medical conditions
* Risk factors for intracranial hemorrhage (trauma, aneurysm, neurosurgery)
* Uncontrolled hypertension or significant coronary or cerebrovascular disease
* Renal or hepatic impairment
* Pregnant, lactating, or of childbearing potential without approved contraception use during ketamine treatment, with a negative urine pregnancy test required at baseline
* Abnormal liver function tests (AST or ALT ≥ 3 times upper normal limit)
* Clinically significant abnormal ECG results
* Unstable thyroid hormone levels or uncorrected hypo or hyper thyroidism
* Any unstable or clinically significant condition judged by the study physician to interfere with treatment
* Positive toxicology screen for drugs not prescribed
* Unwillingness to abstain from benzodiazepines, narcotics, or NMDA antagonists (including memantine and lamotrigine) 12 hours before infusions
* Known intolerance or hypersensitivity to ketamine
* Significant hearing impairment not improved by aids
* Any recent significant decline in exercise tolerance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Study completion AND Adherence to ketamine infusions and ACT psychotherapy sessions | From enrollment to the end of the follow-up at 12 weeks (phase 1, weeks 0 to 12) and from week 1 to week 8
  The number of patients who complete the study (phase 1, weeks 0 to 12). Hypothesis is that at least 80% of enrolled participants will complete the study (week 12 visit).
  The number of patients who complete all ketamine infusions and ACT psychotherapy sessions (weeks 1 to 8). Hypothesis is that at least 80% of enrolled participants will receive at least 75% of all scheduled ketamine infusions and ACT psychotherapy sessions.

SECONDARY OUTCOMES:
Systematic tracking of adverse events and serious adverse events (Safety) | From enrollment to the end of treatment at 8 weeks
  Safety will be assessed through systematic tracking of adverse events (AEs) and serious adverse events (SAEs). AEs occurring during or after ketamine/psychotherapeutic sessions will be solicited and recorded at each study visit according to Medical Dictionary for Regulatory Activities (MedDRA) standards.
  Hypothesis that it will be safe and tolerated, with no SAEs
Recruitment rate | Before enrollment
  The recruitment rate will be calculated as the number of participants enrolled per month. This metric will reflect the feasibility of enrolling eligible individuals within the study timeline. A recruitment rate of 2 to 3 participants per month is anticipated, with full recruitment expected within 10-12 months.
Consent rate | Before enrollment
  The consent rate will represent the proportion of eligible participants who agree to enroll. A consent rate exceeding 80% will be considered indicative of the study's acceptability among the target population.
Data collection rate | From enrollment to the end of treatment at 8 weeks
  The data collection rate will be defined as the proportion of planned data successfully collected across all participants. A rate above 80% will indicate that data collection methods are both feasible and acceptable to participants.
Resource utilization - Therapist | From enrollment to the end of treatment at 8 weeks
  Resource utilization will be systematically tracked throughout the study. For each participant, the following metric will be recorded: therapist time for preparation, delivery, and documentation of ACT sessions. This can help determine whether the intervention is feasible in terms of resource allocation.
Resource utilization - Clinical staff | From enrollment to the end of treatment at 8 weeks
  Resource utilization will be systematically tracked throughout the study. For each participant, the following metric will be recorded: clinical staff time dedicated to ketamine infusions, including nursing, medical monitoring, and recovery supervision. This can help determine whether the intervention is feasible in terms of resource allocation.
Resource utilization - Session duration | From enrollment to the end of treatment at 8 weeks
  Resource utilization will be systematically tracked throughout the study. For each participant, the following metric will be recorded: session duration for both psychotherapy and infusions. This can help determine whether the intervention is feasible in terms of resource allocation.
Resource utilization - Material and infrastructure | From enrollment to the end of treatment at 8 weeks
  Resource utilization will be systematically tracked throughout the study. For each participant, the following metric will be recorded: material and infrastructure use, including room occupancy time, ketamine dosing supplies, monitoring equipment, and music delivery devices. This can help determine whether the intervention is feasible in terms of resource allocation.
Resource utilization - Administrative and coordination time | From enrollment to the end of treatment at 8 weeks
  Resource utilization will be systematically tracked throughout the study. For each participant, the following metric will be recorded: administrative and coordination time, such as scheduling, safety checks (e.g., breathalyzer), and follow-up communication. This can help determine whether the intervention is feasible in terms of resource allocation.
Number of patients engaging in ACT in between therapy exercises | From enrollment to the end of treatment at 8 weeks
  Participant engagement with ACT outside of scheduled therapy sessions will be assessed as a secondary effectiveness measure. This will be defined by the number of between-session exercises completed.

OTHER OUTCOMES:
Change From Baseline in Alcohol Use (TLFB) to End of Treatment and to Follow-up | From enrollment to the end of the follow-up (6 months)
  With the Timeline Followback method, study team provide calendar-based memory cues to help patients build up chronological reports of their alcohol use within an established period. It is considered the gold-standard method to assess alcohol use/quantity.
Change From Baseline in Alcohol Craving (ACQ-NOW) to End of Treatment and to Follow-up | From enrollment to the end of the follow-up (6 months)
  The Alcohol Craving Questionnaire - Now (ACQ-NOW) is a 47-item, self-administered questionnaire designed to assess the intensity and characteristics of alcohol craving at the present moment. Items are rated on a Likert-type scale, and responses are summed to generate a total score, with higher scores indicating greater levels of alcohol craving.
Change From Baseline in Alcohol Craving (OCDS) to End of Treatment and to Follow-up | From enrollment to the end of the follow-up (6 months)
  The Obsessive Compulsive Drinking Scale (OCDS) is a 14-item, self-administered questionnaire designed to assess alcohol related thoughts and behaviors, including obsessive preoccupation with drinking and compulsive drinking behavior. Items are scored using ordinal response options and summed to yield total and subscale scores, with higher scores indicating greater severity of obsessive and compulsive drinking symptoms.
Change From Baseline in SOCRATES (readiness to change alcohol-related behaviors) Total Score to End of Treatment and to Follow-up | From enrollment (baseline) to the end of the follow-up (6 months)
  The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) is a 19-item, self-administered questionnaire designed to assess an individual's readiness to change alcohol related behaviors and engage in treatment. Items are summed to generate total and subscale scores reflecting recognition, ambivalence, and taking steps, with higher scores indicating greater readiness for change and treatment engagement.
Change From Baseline in AASE (self-confidence to avoid alcohol use) Total Score to End of Treatment and to Follow-up | From enrollment (baseline) to the end of the follow-up (6 months)
  The Alcohol Abstinence Self Efficacy Scale (AASE) is a 12-item, self-administered questionnaire designed to assess an individual's confidence in their ability to abstain from alcohol across a range of high risk situations. Items are summed to produce a total score, with higher scores indicating greater abstinence self efficacy.
Change From Baseline in MADRS (depressive symptoms) Total Score to End of Treatment and to Follow-up | From enrollment (baseline) to the end of the follow-up (6 months)
  The Montgomery-Åsberg Depression Rating Scale is a 10-item, clinician-rated scale to rate the severity of the depressive symptoms. Each item is scored from 0 (item's symptoms not present) to 6 (item's symptoms are severe). The total possible score is 60. Higher scores indicate greater severity.
Change From Baseline in BDI-II (depressive symtpoms) Total Score to End of Treatment and to Follow-up | From enrollment (baseline) to the end of the follow-up (6 months)
  The Beck Depression Inventory Scale is a 21-item, patient-rated scale to rate the severity of the depressive symptoms. Each item is scored from 0 (item's symptoms not present) to 3 (item's symptoms are severe). The total possible score is 63. Higher scores indicate greater severity.
Change From Baseline in GAD-7 (general anxiety symptoms) to End of Treatment and Follow-up | From enrollment (baseline) to the end of the follow-up (6 months)
  The General Anxiety Disorder=7 (GAD-7) is a 7 item, self administered measure with scores ranging from 0 to 21, where higher scores indicate worse anxiety symptoms.
Change From Baseline in SSI (suicide ideation) Total to End of Treatment and follow-up | From enrollment (baseline) to the end of the follow-up (6 months)
  The Beck Scale for Suicide Ideation (SSI) is a 19 item, self administered measure with scores ranging from 0 to 38, where higher scores reflect more severe suicide related thoughts.
The Mystical Experience Questionnaire (MEQ) after each ketamine treatment | From the start of ketamine treatment to to the end of ketamine treatment (4 weeks)
  The Mystical Experience Questionnaire consists of 30 statements to rate from 0 (none) to 5 (extreme). Possible scores range from 0 to 150 with higher scores indicating greater mystical experiences.
The Emotional Breakthrough Inventory (EBI) after each ketamine treatment | From the start of ketamine treatment to to the end of ketamine treatment (4 weeks)
  The Emotional Breakthrough Inventory (EBI) is a 6-item, self-administered questionnaire designed to assess the experience of emotional release or breakthrough during psychedelic assisted psychotherapy. Items are rated using Likert-type response options and summed to produce a total score, with higher scores indicating a greater degree of emotional breakthrough.
The Five Facet Mindfulness Questionnaire (FFMQ) at baseline | At enrollment (baseline)
  The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item, self-administered questionnaire designed to assess dispositional mindfulness across five domains, namely observing, describing, acting with awareness, non judging, and non reactivity to inner experience. Items are rated on a Likert-type scale and summed to generate total and facet scores, with higher scores indicating greater levels of mindfulness.
The Modified Tellegen Absorption Scale (MODTAS) at baseline | At enrollment (baseline)
  The Modified Tellegen Absorption Scale (MODTAS) is a 34-item, self-administered questionnaire designed to assess absorption as a personality trait, reflecting an individual's openness to emotional and cognitive alterations across a range of situations. Items are summed to generate a total score, with higher scores indicating greater levels of absorption.
Change From Baseline in EQ-5D-5L (quality of life) to End of Treatment and Follow-up | From enrollment (baseline) to the end of the follow-up (6 months)
  The EQ-5D-5L is a self-administered measure of health related quality of life consisting of two components, a five item descriptive system and a visual analog scale. The descriptive system assesses mobility, self care, usual activities, pain or discomfort, and anxiety or depression, each rated across five levels of severity from no problems to extreme problems. The visual analog scale captures the participant's self rated health on a vertical scale anchored by the worst and best health states imaginable, with higher scores reflecting better perceived health status.
Change From Baseline in WHODAS 2.0 (functioning and disability) to End of Treatment and Follow-up | From enrollment to the end of the follow-up (6 months)
  The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) 12-item version is a self-administered questionnaire designed to assess overall functioning and disability. It evaluates functioning across six domains, including cognition, mobility, self care, interpersonal relationships, daily activities, and social participation. Items are summed to generate an overall functioning score, with higher scores indicating greater levels of disability.
Therapeutic Alliance for participants and for therapists | From the start of psychotherapy treatment to to the end of treatment (8 weeks)
  The Working Alliance Inventory for patient (WAI-SR) is a 12-item, self-administered questionnaire designed to assess the quality of the working alliance between the patient and the therapist. Items evaluate key aspects of the therapeutic alliance and are summed to produce a total score, with higher scores indicating a stronger working alliance. The Working Alliance Inventory - therapist version (WAI-SRT) is a 10-item, self-administered questionnaire completed by the therapist to assess the quality of the working alliance with the patient. Items are summed to yield a total score, with higher scores reflecting a stronger perceived therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Garel, MD MSc, Principal Investigator — Centre Hospitalier d'Université de Montréal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhdanava M, Pilon D, Ghelerter I, Chow W, Joshi K, Lefebvre P, Sheehan JJ. The Prevalence and National Burden of Treatment-Resistant Depression and Major Depressive Disorder in the United States. J Clin Psychiatry. 2021 Mar 16;82(2):20m13699. doi: 10.4088/JCP.20m13699. PMID 33989464
- [Background] Wood E, Bright J, Hsu K, Goel N, Ross JWG, Hanson A, Teed R, Poulin G, Denning B, Corace K, Chase C, Halpape K, Lim R, Kealey T, Rehm J; Canadian Alcohol Use Disorder Guideline Committee. Canadian guideline for the clinical management of high-risk drinking and alcohol use disorder. CMAJ. 2023 Oct 16;195(40):E1364-E1379. doi: 10.1503/cmaj.230715. PMID 37844924
- [Background] Wolff M, Evens R, Mertens LJ, Koslowski M, Betzler F, Grunder G, Jungaberle H. Learning to Let Go: A Cognitive-Behavioral Model of How Psychedelic Therapy Promotes Acceptance. Front Psychiatry. 2020 Feb 21;11:5. doi: 10.3389/fpsyt.2020.00005. eCollection 2020. PMID 32153433
- [Background] Wilkinson ST, Kitay BM, Harper A, Rhee TG, Sint K, Ghosh A, Lopez MO, Saenz S, Tsai J. Barriers to the Implementation of Electroconvulsive Therapy (ECT): Results From a Nationwide Survey of ECT Practitioners. Psychiatr Serv. 2021 Jul 1;72(7):752-757. doi: 10.1176/appi.ps.202000387. Epub 2021 May 11. PMID 33971727
- [Background] Wikberg C, Nejati S, Larsson ME, Petersson EL, Westman J, Ariai N, Kivi M, Eriksson M, Eggertsen R, Hange D, Baigi A, Bjorkelund C. Comparison Between the Montgomery-Asberg Depression Rating Scale-Self and the Beck Depression Inventory II in Primary Care. Prim Care Companion CNS Disord. 2015 Jun 25;17(3):10.4088/PCC.14m01758. doi: 10.4088/PCC.14m01758. eCollection 2015. PMID 26644958
- [Background] Walsh Z, Thiessen MS. Psychedelics and the new behaviourism: considering the integration of third-wave behaviour therapies with psychedelic-assisted therapy. Int Rev Psychiatry. 2018 Aug;30(4):343-349. doi: 10.1080/09540261.2018.1474088. Epub 2018 Sep 25. PMID 30251904
- [Background] Ustun TB, Chatterji S, Kostanjsek N, Rehm J, Kennedy C, Epping-Jordan J, Saxena S, von Korff M, Pull C; WHO/NIH Joint Project. Developing the World Health Organization Disability Assessment Schedule 2.0. Bull World Health Organ. 2010 Nov 1;88(11):815-23. doi: 10.2471/BLT.09.067231. Epub 2010 May 20. PMID 21076562
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] Stubbs KR, Van Bezooyen J, Tang Y-l. Chapter 31 - Managing treatment-resistant depression with comorbid substance use disorders. In: Quevedo J, Riva-Posse P, Bobo WV, editors. Managing Treatment-Resistant Depression: Academic Press; 2022. p. 461-72.
- [Background] Strauss B, Gawlytta R, Schleu A, Frenzl D. Negative effects of psychotherapy: estimating the prevalence in a random national sample. BJPsych Open. 2021;7(6):e186.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Souery D, Oswald P, Massat I, Bailer U, Bollen J, Demyttenaere K, Kasper S, Lecrubier Y, Montgomery S, Serretti A, Zohar J, Mendlewicz J; Group for the Study of Resistant Depression. Clinical factors associated with treatment resistance in major depressive disorder: results from a European multicenter study. J Clin Psychiatry. 2007 Jul;68(7):1062-70. doi: 10.4088/jcp.v68n0713. PMID 17685743
- [Background] Sobell LC, Sobell MB. Timeline Follow-Back. In: Litten RZ, Allen JP, editors. Measuring Alcohol Consumption. Totowa, NJ: Humana Press; 1992. p. 41-72.
- [Background] Smout MF, Longo M, Harrison S, Minniti R, Wickes W, White JM. Psychosocial treatment for methamphetamine use disorders: a preliminary randomized controlled trial of cognitive behavior therapy and Acceptance and Commitment Therapy. Subst Abus. 2010 Apr;31(2):98-107. doi: 10.1080/08897071003641578. PMID 20408061
- [Background] Smith-Apeldoorn SY, Veraart JK, Spijker J, Kamphuis J, Schoevers RA. Maintenance ketamine treatment for depression: a systematic review of efficacy, safety, and tolerability. Lancet Psychiatry. 2022 Nov;9(11):907-921. doi: 10.1016/S2215-0366(22)00317-0. PMID 36244360
- [Background] Sloshower J, Guss J, Krause R, Wallace RM, Williams MT, Reed S, et al. Psilocybin-assisted therapy of major depressive disorder using Acceptance and Commitment Therapy as a therapeutic frame. Journal of Contextual Behavioral Science. 2020;15:12-9.
- [Background] Singleton EG, Gorelick DA. Mechanisms of alcohol craving and their clinical implications. Recent Dev Alcohol. 1998;14:177-95. doi: 10.1007/0-306-47148-5_8. PMID 9751946
- [Background] Singleton E, Tiffany S, Henningfield J. Development and validation of a new questionnaire to assess craving for alcohol. NIDA Research Monograph. 1995;153:289-.
- [Background] Shallcross A, Lu NY, Hays RD. Evaluation of the Psychometric Properties of the Five Facet of Mindfulness Questionnaire. J Psychopathol Behav Assess. 2020 Jun;42(2):271-280. doi: 10.1007/s10862-019-09776-5. Epub 2020 Jan 10. PMID 32655208
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Saunders JB, Aasland OG, Amundsen A, Grant M. Alcohol consumption and related problems among primary health care patients: WHO collaborative project on early detection of persons with harmful alcohol consumption--I. Addiction. 1993 Mar;88(3):349-62. doi: 10.1111/j.1360-0443.1993.tb00822.x. PMID 8461852
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Salani D, Goldin D, Valdes B, DeSantis J. Electroconvulsive Therapy for Treatment-Resistant Depression: Dispelling the Stigma. J Psychosoc Nurs Ment Health Serv. 2023 Jun;61(6):11-17. doi: 10.3928/02793695-20230222-02. Epub 2023 Mar 5. PMID 36853035
- [Background] Sackeim HA. Modern Electroconvulsive Therapy: Vastly Improved yet Greatly Underused. JAMA Psychiatry. 2017 Aug 1;74(8):779-780. doi: 10.1001/jamapsychiatry.2017.1670. No abstract available. PMID 28658461
- [Background] Rothberg RL, Azhari N, Haug NA, Dakwar E. Mystical-type experiences occasioned by ketamine mediate its impact on at-risk drinking: Results from a randomized, controlled trial. J Psychopharmacol. 2021 Feb;35(2):150-158. doi: 10.1177/0269881120970879. Epub 2020 Dec 13. PMID 33307947
- [Background] Roseman L, Haijen E, Idialu-Ikato K, Kaelen M, Watts R, Carhart-Harris R. Emotional breakthrough and psychedelics: Validation of the Emotional Breakthrough Inventory. J Psychopharmacol. 2019 Sep;33(9):1076-1087. doi: 10.1177/0269881119855974. Epub 2019 Jul 11. PMID 31294673
- [Background] Petersen TJ. Enhancing the efficacy of antidepressants with psychotherapy. J Psychopharmacol. 2006 May;20(3 Suppl):19-28. doi: 10.1177/1359786806064314. PMID 16644768
- [Background] Papakostas GI, Thase ME, Fava M, Nelson JC, Shelton RC. Are antidepressant drugs that combine serotonergic and noradrenergic mechanisms of action more effective than the selective serotonin reuptake inhibitors in treating major depressive disorder? A meta-analysis of studies of newer agents. Biol Psychiatry. 2007 Dec 1;62(11):1217-27. doi: 10.1016/j.biopsych.2007.03.027. Epub 2007 Jun 22. PMID 17588546
- [Background] Papakostas GI. Maintaining Rapid Antidepressant Effects Following Ketamine Infusion: A Major Unmet Need. J Clin Psychiatry. 2020 Feb 4;81(2):19r12859. doi: 10.4088/JCP.19r12859. PMID 32023369
- [Background] Pahnke WN. Psychedelic drugs and mystical experience. Int Psychiatry Clin. 1969;5(4):149-62. No abstract available. PMID 4892137
- [Background] Pahnke WN. Drugs and Mysticism: An Analysis of the Relationship Between Psychedelic Drugs and the Mystical Consciousness : a Thesis: Harvard University; 1963.
- [Background] Osaji J, Ojimba C, Ahmed S. The Use of Acceptance and Commitment Therapy in Substance Use Disorders: A Review of Literature. J Clin Med Res. 2020 Oct;12(10):629-633. doi: 10.14740/jocmr4311. Epub 2020 Sep 21. PMID 33029268
- [Background] Oliveira-Maia AJ, Bobrowska A, Constant E, Ito T, Kambarov Y, Luedke H, Mulhern-Haughey S, von Holt C. Treatment-Resistant Depression in Real-World Clinical Practice: A Systematic Literature Review of Data from 2012 to 2022. Adv Ther. 2024 Jan;41(1):34-64. doi: 10.1007/s12325-023-02700-0. Epub 2023 Oct 26. PMID 37882883
- [Background] Nikolin S, Rodgers A, Schwaab A, Bahji A, Zarate C Jr, Vazquez G, Loo C. Ketamine for the treatment of major depression: a systematic review and meta-analysis. EClinicalMedicine. 2023 Aug 3;62:102127. doi: 10.1016/j.eclinm.2023.102127. eCollection 2023 Aug. PMID 37593223
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Mollaahmetoglu OM, Keeler J, Ashbullby KJ, Ketzitzidou-Argyri E, Grabski M, Morgan CJA. "This Is Something That Changed My Life": A Qualitative Study of Patients' Experiences in a Clinical Trial of Ketamine Treatment for Alcohol Use Disorders. Front Psychiatry. 2021 Aug 16;12:695335. doi: 10.3389/fpsyt.2021.695335. eCollection 2021. PMID 34483991
- [Background] Meis LA, Griffin JM, Greer N, Jensen AC, Macdonald R, Carlyle M, Rutks I, Wilt TJ. Couple and family involvement in adult mental health treatment: a systematic review. Clin Psychol Rev. 2013 Mar;33(2):275-86. doi: 10.1016/j.cpr.2012.12.003. Epub 2012 Dec 22. PMID 23321286
- [Background] McPheeters M, O'Connor EA, Riley S, Kennedy SM, Voisin C, Kuznacic K, Coffey CP, Edlund MD, Bobashev G, Jonas DE. Pharmacotherapy for Alcohol Use Disorder: A Systematic Review and Meta-Analysis. JAMA. 2023 Nov 7;330(17):1653-1665. doi: 10.1001/jama.2023.19761. PMID 37934220
- [Background] McMullen EP, Lee Y, Lipsitz O, Lui LMW, Vinberg M, Ho R, Rodrigues NB, Rosenblat JD, Cao B, Gill H, Teopiz KM, Cha DS, McIntyre RS. Strategies to Prolong Ketamine's Efficacy in Adults with Treatment-Resistant Depression. Adv Ther. 2021 Jun;38(6):2795-2820. doi: 10.1007/s12325-021-01732-8. Epub 2021 Apr 30. PMID 33929660
- [Background] McKiernan P, Cloud R, Patterson DA, Wolf Adelv Unegv Waya S, Golder S, Besel K. Development of a Brief Abstinence Self-Efficacy Measure. J Soc Work Pract Addict. 2011 Jul;11(3):245-253. doi: 10.1080/1533256X.2011.593445. Epub 2011 Aug 16. PMID 23559892
- [Background] McIntyre RS, Alsuwaidan M, Baune BT, Berk M, Demyttenaere K, Goldberg JF, Gorwood P, Ho R, Kasper S, Kennedy SH, Ly-Uson J, Mansur RB, McAllister-Williams RH, Murrough JW, Nemeroff CB, Nierenberg AA, Rosenblat JD, Sanacora G, Schatzberg AF, Shelton R, Stahl SM, Trivedi MH, Vieta E, Vinberg M, Williams N, Young AH, Maj M. Treatment-resistant depression: definition, prevalence, detection, management, and investigational interventions. World Psychiatry. 2023 Oct;22(3):394-412. doi: 10.1002/wps.21120. PMID 37713549
- [Background] McHugh RK, Weiss RD. Alcohol Use Disorder and Depressive Disorders. Alcohol Res. 2019 Jan 1;40(1):arcr.v40.1.01. doi: 10.35946/arcr.v40.1.01. eCollection 2019 Oct 21. PMID 31649834
- [Background] Mathai DS, Mora V, Garcia-Romeu A. Toward Synergies of Ketamine and Psychotherapy. Front Psychol. 2022 Mar 25;13:868103. doi: 10.3389/fpsyg.2022.868103. eCollection 2022. PMID 35401323
- [Background] Marini C, Northover NS, Gold ND, Rogers UK, O'Donnell KC, Tofighi B, Ross S, Bogenschutz MP. A Systematic Approach to Standardizing Drinking Outcomes From Timeline Followback Data. Subst Abuse. 2023 Mar 11;17:11782218231157558. doi: 10.1177/11782218231157558. eCollection 2023. PMID 36923069
- [Background] Magill M, Ray L, Kiluk B, Hoadley A, Bernstein M, Tonigan JS, Carroll K. A meta-analysis of cognitive-behavioral therapy for alcohol or other drug use disorders: Treatment efficacy by contrast condition. J Consult Clin Psychol. 2019 Dec;87(12):1093-1105. doi: 10.1037/ccp0000447. Epub 2019 Oct 10. PMID 31599606
- [Background] MacLeod MA, Tremblay PF, Graham K, Bernards S, Rehm J, Wells S. Psychometric properties and a latent class analysis of the 12-item World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) in a pooled dataset of community samples. Int J Methods Psychiatr Res. 2016 Dec;25(4):243-254. doi: 10.1002/mpr.1523. Epub 2016 Sep 15. PMID 27634553
- [Background] Maclean KA, Leoutsakos JM, Johnson MW, Griffiths RR. Factor Analysis of the Mystical Experience Questionnaire: A Study of Experiences Occasioned by the Hallucinogen Psilocybin. J Sci Study Relig. 2012 Dec;51(4):721-737. doi: 10.1111/j.1468-5906.2012.01685.x. PMID 23316089
- [Background] Lee EB, An W, Levin ME, Twohig MP. An initial meta-analysis of Acceptance and Commitment Therapy for treating substance use disorders. Drug Alcohol Depend. 2015 Oct 1;155:1-7. doi: 10.1016/j.drugalcdep.2015.08.004. Epub 2015 Aug 13. PMID 26298552
- [Background] Krystal JH, Abdallah CG, Sanacora G, Charney DS, Duman RS. Ketamine: A Paradigm Shift for Depression Research and Treatment. Neuron. 2019 Mar 6;101(5):774-778. doi: 10.1016/j.neuron.2019.02.005. PMID 30844397
- [Background] Kryst J, Kawalec P, Mitoraj AM, Pilc A, Lason W, Brzostek T. Efficacy of single and repeated administration of ketamine in unipolar and bipolar depression: a meta-analysis of randomized clinical trials. Pharmacol Rep. 2020 Jun;72(3):543-562. doi: 10.1007/s43440-020-00097-z. Epub 2020 Apr 16. PMID 32301056
- [Background] Kranzler HR, Soyka M. Diagnosis and Pharmacotherapy of Alcohol Use Disorder: A Review. JAMA. 2018 Aug 28;320(8):815-824. doi: 10.1001/jama.2018.11406. PMID 30167705
- [Background] Koob GF. Alcohol Use Disorder Treatment: Problems and Solutions. Annu Rev Pharmacol Toxicol. 2024 Jan 23;64:255-275. doi: 10.1146/annurev-pharmtox-031323-115847. PMID 38261428
- [Background] Klein JP, Rozental A, Surig S, Moritz S. Adverse Events of Psychological Interventions: Definitions, Assessment, Current State of the Research and Implications for Research and Clinical Practice. Psychother Psychosom. 2024;93(5):308-315. doi: 10.1159/000540212. Epub 2024 Jul 29. PMID 39074446
- [Background] Klatte R, Strauss B, Fluckiger C, Rosendahl J. Adverse events in psychotherapy randomized controlled trials: A systematic review. Psychother Res. 2025 Jan;35(1):84-99. doi: 10.1080/10503307.2023.2286992. Epub 2023 Dec 13. PMID 38090772
- [Background] Kang MJY, Hawken E, Vazquez GH. The Mechanisms Behind Rapid Antidepressant Effects of Ketamine: A Systematic Review With a Focus on Molecular Neuroplasticity. Front Psychiatry. 2022 Apr 25;13:860882. doi: 10.3389/fpsyt.2022.860882. eCollection 2022. PMID 35546951
- [Background] Jonas DE, Amick HR, Feltner C, Bobashev G, Thomas K, Wines R, Kim MM, Shanahan E, Gass CE, Rowe CJ, Garbutt JC. Pharmacotherapy for adults with alcohol use disorders in outpatient settings: a systematic review and meta-analysis. JAMA. 2014 May 14;311(18):1889-900. doi: 10.1001/jama.2014.3628. PMID 24825644
- [Background] Jimenez M, Grana JL, Montes V, Rubio G. Alcohol craving scale based on three factors. Eur Addict Res. 2009;15(3):135-42. doi: 10.1159/000210043. Epub 2009 Mar 31. PMID 19332992
- [Background] Hunt GE, Malhi GS, Lai HMX, Cleary M. Prevalence of comorbid substance use in major depressive disorder in community and clinical settings, 1990-2019: Systematic review and meta-analysis. J Affect Disord. 2020 Apr 1;266:288-304. doi: 10.1016/j.jad.2020.01.141. Epub 2020 Jan 26. PMID 32056890
- [Background] Hoeppner BB, Stout RL, Jackson KM, Barnett NP. How good is fine-grained Timeline Follow-back data? Comparing 30-day TLFB and repeated 7-day TLFB alcohol consumption reports on the person and daily level. Addict Behav. 2010 Dec;35(12):1138-43. doi: 10.1016/j.addbeh.2010.08.013. Epub 2010 Aug 13. PMID 20822852
- [Background] Higgins-Biddle JC, Babor TF. A review of the Alcohol Use Disorders Identification Test (AUDIT), AUDIT-C, and USAUDIT for screening in the United States: Past issues and future directions. Am J Drug Alcohol Abuse. 2018;44(6):578-586. doi: 10.1080/00952990.2018.1456545. Epub 2018 May 3. PMID 29723083
- [Background] Hermida AP, Glass OM, Shafi H, McDonald WM. Electroconvulsive Therapy in Depression: Current Practice and Future Direction. Psychiatr Clin North Am. 2018 Sep;41(3):341-353. doi: 10.1016/j.psc.2018.04.001. Epub 2018 Jun 15. PMID 30098649
- [Background] Henssler J, Kurschus M, Franklin J, Bschor T, Baethge C. Trajectories of Acute Antidepressant Efficacy: How Long to Wait for Response? A Systematic Review and Meta-Analysis of Long-Term, Placebo-Controlled Acute Treatment Trials. J Clin Psychiatry. 2018 May/Jun;79(3):17r11470. doi: 10.4088/JCP.17r11470. PMID 29659207
- [Background] Henssler J, Alexander D, Schwarzer G, Bschor T, Baethge C. Combining Antidepressants vs Antidepressant Monotherapy for Treatment of Patients With Acute Depression: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2022 Apr 1;79(4):300-312. doi: 10.1001/jamapsychiatry.2021.4313. PMID 35171215
- [Background] Heerlein K, Perugi G, Otte C, Frodl T, Degraeve G, Hagedoorn W, Oliveira-Maia AJ, Perez Sola V, Rathod S, Rosso G, Sierra P, Malynn S, Morrens J, Verrijcken C, Gonzalez B, Young AH. Real-world evidence from a European cohort study of patients with treatment resistant depression: Treatment patterns and clinical outcomes. J Affect Disord. 2021 Jul 1;290:334-344. doi: 10.1016/j.jad.2021.03.073. Epub 2021 Apr 1. PMID 34044256
- [Background] Hayes SC, Wilson KG, Gifford EV, Bissett R, Piasecki M, Batten SV, et al. A Preliminary trial of twelve-step facilitation and acceptance and commitment therapy with polysubstance-abusing methadone-maintained opiate addicts. Behavior Therapy. 2004;35(4):667-88.
- [Background] Hasin DS, Wall M, Witkiewitz K, Kranzler HR, Falk D, Litten R, Mann K, O'Malley SS, Scodes J, Robinson RL, Anton R; Alcohol Clinical Trials Initiative (ACTIVE) Workgroup. Change in non-abstinent WHO drinking risk levels and alcohol dependence: a 3 year follow-up study in the US general population. Lancet Psychiatry. 2017 Jun;4(6):469-476. doi: 10.1016/S2215-0366(17)30130-X. Epub 2017 Apr 26. PMID 28456501
- [Background] Hasin DS, Sarvet AL, Meyers JL, Saha TD, Ruan WJ, Stohl M, Grant BF. Epidemiology of Adult DSM-5 Major Depressive Disorder and Its Specifiers in the United States. JAMA Psychiatry. 2018 Apr 1;75(4):336-346. doi: 10.1001/jamapsychiatry.2017.4602. PMID 29450462
- [Background] Hall W, Saunders JB, Babor TF, Aasland OG, Amundsen A, Hodgson R, Grant M. The structure and correlates of alcohol dependence: WHO collaborative project on the early detection of persons with harmful alcohol consumption--III. Addiction. 1993 Dec;88(12):1627-36. doi: 10.1111/j.1360-0443.1993.tb02037.x. PMID 7907509
- [Background] Grant S, Azhar G, Han E, Booth M, Motala A, Larkin J, Hempel S. Clinical interventions for adults with comorbid alcohol use and depressive disorders: A systematic review and network meta-analysis. PLoS Med. 2021 Oct 8;18(10):e1003822. doi: 10.1371/journal.pmed.1003822. eCollection 2021 Oct. PMID 34624018
- [Background] Grant BF, Goldstein RB, Saha TD, Chou SP, Jung J, Zhang H, Pickering RP, Ruan WJ, Smith SM, Huang B, Hasin DS. Epidemiology of DSM-5 Alcohol Use Disorder: Results From the National Epidemiologic Survey on Alcohol and Related Conditions III. JAMA Psychiatry. 2015 Aug;72(8):757-66. doi: 10.1001/jamapsychiatry.2015.0584. PMID 26039070
- [Background] Grabski M, McAndrew A, Lawn W, Marsh B, Raymen L, Stevens T, Hardy L, Warren F, Bloomfield M, Borissova A, Maschauer E, Broomby R, Price R, Coathup R, Gilhooly D, Palmer E, Gordon-Williams R, Hill R, Harris J, Mollaahmetoglu OM, Curran HV, Brandner B, Lingford-Hughes A, Morgan CJA. Adjunctive Ketamine With Relapse Prevention-Based Psychological Therapy in the Treatment of Alcohol Use Disorder. Am J Psychiatry. 2022 Feb;179(2):152-162. doi: 10.1176/appi.ajp.2021.21030277. Epub 2022 Jan 11. PMID 35012326
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Felton JW, Strutz KL, McCauley HL, Poland CA, Barnhart KJ, Lejuez CW. Delay Discounting Interacts with Distress Tolerance to Predict Depression and Alcohol Use Disorders among Individuals Receiving Inpatient Substance Use Services. Int J Ment Health Addict. 2020 Oct;18(5):1416-1421. doi: 10.1007/s11469-019-00163-5. Epub 2019 Nov 14. PMID 33312085
- [Background] Espinoza RT, Kellner CH. Electroconvulsive Therapy. N Engl J Med. 2022 Feb 17;386(7):667-672. doi: 10.1056/NEJMra2034954. No abstract available. PMID 35172057
- [Background] DiClemente CC, Carbonari JP, Montgomery RP, Hughes SO. The Alcohol Abstinence Self-Efficacy scale. J Stud Alcohol. 1994 Mar;55(2):141-8. doi: 10.15288/jsa.1994.55.141. PMID 8189734
- [Background] Devlin N, Pickard S, Busschbach J. The Development of the EQ-5D-5L and its Value Sets. In: Devlin N, Roudijk B, Ludwig K, editors. Value Sets for EQ-5D-5L: A Compendium, Comparative Review &amp;amp;amp;amp; User Guide. Cham (CH): Springer Copyright 2022, The Author(s). 2022. p. 1-12.
- [Background] de Jonghe F, Kool S, van Aalst G, Dekker J, Peen J. Combining psychotherapy and antidepressants in the treatment of depression. J Affect Disord. 2001 May;64(2-3):217-29. doi: 10.1016/s0165-0327(00)00259-7. PMID 11313088
- [Background] Davis AK, Barrett FS, Griffiths RR. Psychological flexibility mediates the relations between acute psychedelic effects and subjective decreases in depression and anxiety. J Contextual Behav Sci. 2020 Jan;15:39-45. doi: 10.1016/j.jcbs.2019.11.004. Epub 2019 Nov 16. PMID 32864325
- [Background] Davidson J, Turnbull CD, Strickland R, Miller R, Graves K. The Montgomery-Asberg Depression Scale: reliability and validity. Acta Psychiatr Scand. 1986 May;73(5):544-8. doi: 10.1111/j.1600-0447.1986.tb02723.x. PMID 3751660
- [Background] Das RK, Gale G, Walsh K, Hennessy VE, Iskandar G, Mordecai LA, Brandner B, Kindt M, Curran HV, Kamboj SK. Ketamine can reduce harmful drinking by pharmacologically rewriting drinking memories. Nat Commun. 2019 Nov 26;10(1):5187. doi: 10.1038/s41467-019-13162-w. PMID 31772157
- [Background] Dakwar E, Levin F, Hart CL, Basaraba C, Choi J, Pavlicova M, Nunes EV. A Single Ketamine Infusion Combined With Motivational Enhancement Therapy for Alcohol Use Disorder: A Randomized Midazolam-Controlled Pilot Trial. Am J Psychiatry. 2020 Feb 1;177(2):125-133. doi: 10.1176/appi.ajp.2019.19070684. Epub 2019 Dec 2. PMID 31786934
- [Background] Craighead WE, Dunlop BW. Combination psychotherapy and antidepressant medication treatment for depression: for whom, when, and how. Annu Rev Psychol. 2014;65:267-300. doi: 10.1146/annurev.psych.121208.131653. Epub 2013 Sep 13. PMID 24405361
- [Background] Conigrave KM, Hall WD, Saunders JB. The AUDIT questionnaire: choosing a cut-off score. Alcohol Use Disorder Identification Test. Addiction. 1995 Oct;90(10):1349-56. doi: 10.1046/j.1360-0443.1995.901013496.x. PMID 8616463
- [Background] Close JB, Hajien EC, Watts R, Roseman L, Carhart-Harris RL. Psychedelics and psychological flexibility - Results of a prospective web-survey using the Acceptance and Action Questionnaire II. Journal of Contextual Behavioral Science. 2020;16:37-44.
- [Background] Carvalho AF, Heilig M, Perez A, Probst C, Rehm J. Alcohol use disorders. Lancet. 2019 Aug 31;394(10200):781-792. doi: 10.1016/S0140-6736(19)31775-1. PMID 31478502
- [Background] Bschor T, Kern H, Henssler J, Baethge C. Switching the Antidepressant After Nonresponse in Adults With Major Depression: A Systematic Literature Search and Meta-Analysis. J Clin Psychiatry. 2018 Jan/Feb;79(1):16r10749. doi: 10.4088/JCP.16r10749. PMID 27929611
- [Background] Brenner P, Brandt L, Li G, DiBernardo A, Boden R, Reutfors J. Substance use disorders and risk for treatment resistant depression: a population-based, nested case-control study. Addiction. 2020 Apr;115(4):768-777. doi: 10.1111/add.14866. Epub 2019 Dec 16. PMID 31656053
- [Background] Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): validation of a screening instrument for use in medical settings. J Stud Alcohol. 1995 Jul;56(4):423-32. doi: 10.15288/jsa.1995.56.423. PMID 7674678
- [Background] Bilbao A, Martin-Fernandez J, Garcia-Perez L, Mendezona JI, Arrasate M, Candela R, Acosta FJ, Estebanez S, Retolaza A. Psychometric properties of the EQ-5D-5L in patients with major depression: factor analysis and Rasch analysis. J Ment Health. 2022 Aug;31(4):506-516. doi: 10.1080/09638237.2021.1875422. Epub 2021 Feb 1. PMID 33522336
- [Background] Bernstein EY, Baggett TP, Trivedi S, Herzig SJ, Anderson TS. Pharmacologic Treatment Initiation Among Medicare Beneficiaries Hospitalized With Alcohol Use Disorder. Ann Intern Med. 2023 Aug;176(8):1137-1139. doi: 10.7326/M23-0641. Epub 2023 Jun 27. No abstract available. PMID 37364264
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Anton RF, Moak DH, Latham PK. The obsessive compulsive drinking scale: A new method of assessing outcome in alcoholism treatment studies. Arch Gen Psychiatry. 1996 Mar;53(3):225-31. doi: 10.1001/archpsyc.1996.01830030047008. PMID 8611059
- [Background] Anton RF, Moak DH, Latham P. The Obsessive Compulsive Drinking Scale: a self-rated instrument for the quantification of thoughts about alcohol and drinking behavior. Alcohol Clin Exp Res. 1995 Feb;19(1):92-9. doi: 10.1111/j.1530-0277.1995.tb01475.x. PMID 7771669
- [Background] Anand A, Mathew SJ, Sanacora G, Murrough JW, Goes FS, Altinay M, Aloysi AS, Asghar-Ali AA, Barnett BS, Chang LC, Collins KA, Costi S, Iqbal S, Jha MK, Krishnan K, Malone DA, Nikayin S, Nissen SE, Ostroff RB, Reti IM, Wilkinson ST, Wolski K, Hu B. Ketamine versus ECT for Nonpsychotic Treatment-Resistant Major Depression. N Engl J Med. 2023 Jun 22;388(25):2315-2325. doi: 10.1056/NEJMoa2302399. Epub 2023 May 24. PMID 37224232
- [Background] Alsheikh AM, Elemam MO, El-Bahnasawi M. Treatment of Depression With Alcohol and Substance Dependence: A Systematic Review. Cureus. 2020 Oct 26;12(10):e11168. doi: 10.7759/cureus.11168. PMID 33133799
- [Background] Alnefeesi Y, Chen-Li D, Krane E, Jawad MY, Rodrigues NB, Ceban F, Di Vincenzo JD, Meshkat S, Ho RCM, Gill H, Teopiz KM, Cao B, Lee Y, McIntyre RS, Rosenblat JD. Real-world effectiveness of ketamine in treatment-resistant depression: A systematic review & meta-analysis. J Psychiatr Res. 2022 Jul;151:693-709. doi: 10.1016/j.jpsychires.2022.04.037. Epub 2022 May 25. PMID 35688035
- [Background] Allen JP, Litten RZ, Fertig JB, Babor T. A review of research on the Alcohol Use Disorders Identification Test (AUDIT). Alcohol Clin Exp Res. 1997 Jun;21(4):613-9. PMID 9194913